CLINICAL TRIAL: NCT02113254
Title: Study of Modification of the Density of the Macular Pigment by the Consumption of Corn With Strong Content in Zeaxanthine
Brief Title: Study of the Macular Pigment by the Consumption of Corn With Strong Content in Zeaxanthine
Acronym: MAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Vilmorin & Cie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2013/17
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Age Macular Degeneration
Keywords: corn; macular pigment; lutein; zeaxanthin; Age Macular Degeneration; AMD
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteer (Experimental)
  Interventions: Other: Corn zeaxanthin

INTERVENTIONS:
Other: Corn zeaxanthin — The treatment will consist in a daily consumption of a box of 125g of corn with strong zeaxanthin content during 10 weeks. This corresponds to a daily contribution of at least 1,2 mg of lutein and 2,2 mg de zeaxanthin

SUMMARY:
The Age Macular Degeneration (AMD) is the first cause of blindness in industrialized countries. The macular pigment (lutein and zeaxanthin) could play an important role in the arisen of the AMD. The food supplementation by corn with strong concentration in macular pigment could increase the density of the macular pigment. This could, in the future, represent a strategy of prevention of the AMD. The main objective of this study is to detect an increase of the macular pigment density after the consumption of this corn at healthy volunteers.

DETAILED DESCRIPTION:
The age macular degeneration represents the first cause of blindness in industrialized countries if it is not treated. In France, the AMD affects 600 000 persons and this figure should continue to increase, notably because of the increase of the life expectancy. The macula is responsible of the fine vision, the vision of colours and the perception of contrasts. The macular pigment is present only at the level of the macular area. This pigment is composed of three carotenoids: lutein, zeaxanthin, meso-zeaxanthin. The first two compounds are of strictly food origin and are not produced in an endogenous way. A change of the macular pigment density and/or the quality of the macular pigment is suspected to play a role in the appearance and the evolution of the AMD. The food supplementation by corn with strong concentration in macular pigment could increase the density of the macular pigment. This could, in the future, represent a strategy of prevention of the AMD. The main objective of this study is to detect an increase of the macular pigment density after the consumption of this corn at healthy volunteers. The treatment will consist in a daily consumption of a box of 125g of corn with strong zeaxanthin content during 10 weeks. This corresponds to a daily contribution of at least 1,2 mg of lutein and 2,2 mg de zeaxanthin. After the inclusion visit, the subject will be seen 5 times (after 3, 6, 8, 10, 14 weeks of treatment). In all these visits, measures of the macular pigment will be realized. A blood sample will be realized at the inclusion visit and during the visit at 6 and 10 weeks.

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteers, men and women
* Corrected visual acuity upper or equal to 8/10 in two eyes.
* Age: 20 - 35 years
* Free and written consent signed by the participant and the investigator before any examination required by the research
* Subject agreeing to be registered in the national file
* Affiliated subject of a national insurance scheme

Exclusion criteria:

* Presence of AMD signs on one or two eyes
* Histories of other evolutionary ocular pathologies susceptible to complicate the evaluation of the AMD and of the visual acuity (glaucoma, high myopia forte (>= - 6 dioptres), strong retinopathy…)
* Subject operated of de cataract
* Lens Opacities (NO>=3, et/ou NC>=3, et/ou C>=1 et/ou P>=1 according to the LOCSII method)
* Food complements in the year wich precedes (list of complements in appendix 2)
* Hypersensitive people in the tropicamide, in the atropine, its by-products, or in one of the excipients of the tropicamide
* Patients at risk of angle closure glaucoma
* Body Masse Index >= 30 kg/m2
* Current smoking or stop for less than 12 months
* Diabetes
* High blood pressure
* Hyperlipidemia
* Neuro-inflammatory diseases
* Chronical gastro-intestinal diseases (Crohn …)
* Taking of continuous medicine during more than one month, during the last 12 months (exception of the contraceptive pill)
* Pregnant or breast-feeding woman
* Vegetarian Patient
* Participation in another clinical trial during 30 days wich precedes
* Not compliant subjects
* Subject without french national insurance scheme
* Subject under guardianship judicial

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the measure of the evolution of the macular pigment density after 10 weeks of supplementation compared with the initial measure. | 10 weeks after inclusion

SECONDARY OUTCOMES:
The measure of the evolution of the plasmatic rate of zeaxanthin after10 weeks of supplementation | 10 weeks after inclusion
The measure of the macular pigment density before supplementation in 3, 6, 8, and 10 weeks of supplementation and after 4 weeks of stop by three methods: the sensibility in colours and two methods of autofluorescence | 10 weeks after inclusion
The measure of plasmatic rate of total cholesterol, HDL-cholesterol, triglycerides, lutein and zeaxanthin, initial and in 6 and 10 weeks of supplementation | 10 weeks after inclusion
In the inclusion, the measure of the visual acuity and the examination of the fundus oculi. | 10 weeks after inclusion
In the inclusion, the measure of the retinal thickness with OCT (Optical Coherence Tomography) | 10 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François KOROBELNIK, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France